CLINICAL TRIAL: NCT03779581
Title: Self Correction Exercises for Idiopathic Scoliosis Among Adolescents
Brief Title: Self Correction Exercises for Idiopathic Scoliosis Among Adolescents. A Randomised Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Lecturer, Department of physical Therapy and Health Rehabilitation, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MajmaahUniversity
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Scoliosis Idiopathic
MeSH Terms: interventions — Orthotic Devices

STUDY DESIGN:
Intervention Model Description: 1431 of the 108 subjects visiting out-patient Department of our hospital met the inclusion criteria. All the subjects diagnosed with kyphoscoliosis signed the informed consent approved by the ethical committee of the hospital. The diagnosis was based on the diagnosis by an experienced radiologist. Subjects with idiopathic kyphoscoliosis and Cobb's angle greater than 60 degree and normal pulmonary function were included. The subjects with other cardiovascular pathologies, congenital disorders and inability to commute were excluded from this study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The researcher, surgeons, and physiotherapist did not participate in randomization, treatment, or outcome assessments. The assessor was blinded. A computer-generated sequence inside pre-sealed opaque envelopes with sequentially numbered opaque envelopes randomly allocated individuals to the groups. To ensure a fair distribution of curve types between the two groups (54 per group), a random size (4-8) blocked randomization was stratified for the six curve types. Participants were asked not to reveal their group affiliations to ensure evaluators were blind. The statistician was also insulated from group allocation coding. During routine clinic visits, a trained technician blinded to study participation took radiographs. An expert blinded to groups and time measured the radiographs.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): The experimental group received active self-correction exercises to restore movements in different planes as close as possible to physiologically normal.
  Interventions: Other: Self Correction exercises
- Control Group (Active Comparator): All patients were prescribed a spinal orthosis (TLSO) and got a preliminary evaluation for orthosis design and manufacturing based on the curve type categorization from Ross and Weiss during the first appointment (Rigo et al., 2010).
  Interventions: Device: orthotic devices

INTERVENTIONS:
Other: Self Correction exercises — Active self-correction exercises to restore movements in different planes as close to physiologically normal as possible.
  Arms: Exercise Group
Device: orthotic devices — the orthotic devices designed to correct the scoliosis curve
  Arms: Control Group

SUMMARY:
Adolescent idiopathic scoliosis (AIS) is a three-dimensional spinal deformity with an unknown cause that affects adolescents aged 10 or older. A standing posterior-anterior radiograph with a Cobb angle greater than 10 degrees is used to make the diagnosis. Depending on the severity of the spinal deformity, conservative treatments and surgery are used to treat AIS. Patients whose spinal curvature is greater than 45 degrees are typically considered for surgery. The majority of patients with AIS receive conservative treatments to prevent and slow the progression of the curve. 2 Orthotic intervention (OI) and scoliosis-specific exercise (SSE) are commonly recommended by the International Society on Scoliosis Orthopaedic and Rehabilitation Treatment for patients with a curvature between 20 and 45 degrees. Self correction exercises are the group of spinal extension, lateral spinal flexion and rotational exercises performed to correct spinal deviation. Exercises are performed in a different fundamental postures.

DETAILED DESCRIPTION:
Scoliosis is a malformation of the musculoskeletal system that is defined by lateral deviation of the spine, which is typically accompanied by vertebral rotation and lordosis. The term "scoliosis" refers to the curvature of the spine that results from the condition (3-dimensional deformity). Scoliosis in female teenagers often reaches its most advanced stage between the ages of 11 and 16 years old. In general, scoliosis may be broken down into two categories: structural and non-structural scoliosis. The level of severity and the degree of deformity of the spine are the major characteristics that differentiate the two groups. It is common practice to refer to the structural type of scoliosis as a sort of spinal deformity that cannot be corrected without surgical intervention. Bracing, exercises, and education are some of the conservative treatments that may be used to control non-structural spinal deformity, which is a movable disorder. Scoliosis that is not treated properly may advance to a functionally degraded condition, which is characterized by physical asymmetry, muscular imbalance, back discomfort, and considerable respiratory disruption. This can lead to distorted body image and a loss of self-esteem in the patient. Idiopathic adolescent scoliosis, more commonly known as AIS, is the diagnosis that is typically made in children who are otherwise healthy but have a spinal curvature of at least ten degrees but less than fifty degrees. This curvature range is what determines whether a child is considered to have AIS. While treating scoliosis, the primary goal of therapy should be to slow or stop the disease's development so that the treatment may be regarded effective. Non-conservative therapies often entail surgical techniques for the correction of spinal abnormalities; nevertheless, these operations do not come without associated risks. Individuals who arrive with a scoliosis curvature of less than 40 degrees have the potential to be candidates for conservative treatments such as physiotherapy scoliosis-specific exercise (PSSE), with or without the concomitant use of an external brace.

ELIGIBILITY:
10-16-year-olds with AIS, all sexes, all curve kinds, curves between 10° and 45°, Risser grade 0 to 5, with or without brace, and the capacity to attend weekly checkups.

Exclusion criteria included patients with a diagnosis other than AIS, those who had finished brace therapy, those planned for surgery, those with a follow-up scheduled beyond 62 months, and those who had had prior spine surgery.

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Cobb angle | 1-2 hours
  Angulation calculated on X-ray
SRS 22 | 1-2 hours
  Scoliosis rating scale 22 items

CONTACTS AND LOCATIONS:
Locations (1):
- Faizan Kashoo, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided